CLINICAL TRIAL: NCT06881043
Title: A Multicenter, Prospective, Observational Cohort Study to Assess the Safety and Efficacy of Robotic Assisted Surgery Using Vessel Sealer Extend in Locally Advanced Gastric Cancer (STARS-GC09)
Brief Title: The Safety and Efficacy of Robotic Assisted Surgery Using Vessel Sealer Extend in Locally Advanced Gastric Cancer
Acronym: STARS-GC09
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); The First Affiliated Hospital of Soochow University (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Quan Wang, Director, Clinical Professor, The First Hospital of Jilin University
Other Study IDs: STARS-GC09
Record Dates: First submitted 2025-03-03; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Gastric Cancer; Gastric Adenocarcinoma
Keywords: Robot-assisted surgery; Vessel sealer extend; Gastrectomy; Laparoscopic-assisted surgery; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Robot-assisted radical gastrectomy using VSE for locally advanced gastric cancer.: The surgeon performed robot-assisted radical gastrectomy using VSE for locally advanced gastric cancer.
- laparoscopic-assisted radical gastrectomy for advanced gastric cancer: The surgeon performed laparoscopic-assisted radical gastrectomy for advanced gastric cancer.

SUMMARY:
Gastric cancer is the fifth most common malignancy and the fourth leading cause of cancer-related deaths. Surgical resection is the primary treatment, with laparoscopic-assisted gastrectomy (LG) being a minimally invasive option. However, LG is limited by restricted instrument mobility and hand tremors, which affect precision. The Da Vinci robotic system enhances surgical precision with 3D magnification, improved hand-eye coordination, tremor filtration, and flexible instruments. It is especially beneficial in complex procedures like D2 lymph node dissection and lower mediastinal lymph node clearance. Unlike laparoscopic surgery, robotic surgery offers superior flexibility and reduced pancreatic injury during dissection. Robotic-assisted gastrectomy (RG) offers advantages over LG, such as reduced blood loss, shorter hospital stays, and improved lymph node dissection. However, its short-term benefits remain debated, and most studies focus on early gastric cancer. The safety and efficacy of RG for advanced gastric cancer are not well-established.

Vascular coagulation is crucial in minimally invasive surgery. Ultrasonic devices, though widely used, can cause thermal damage due to high temperatures. In contrast, the Vessel Sealer Extend (VSE) offers greater flexibility and precision. It allows 540° instrument rotation, coagulates vessels up to 7 mm in diameter with lower energy, and minimizes thermal injury. Retrospective studies show RG with VSE may have faster recovery and fewer complications than LG. However, further prospective, multicenter studies are needed to confirm these benefits for advanced gastric cancer.

The investigators propose a multicenter, observational study to evaluate RG with VSE in advanced gastric cancer, assessing safety, recovery, and oncological outcomes.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common malignancy worldwide and the fourth leading cause of cancer-related deaths. Surgical resection remains the primary treatment for the radical management of gastric cancer. Laparoscopic-assisted gastrectomy (LG) has proven to be a minimally invasive and safe approach for both early-stage and advanced gastric cancer, offering significant advantages over open surgery. However, LG is still limited by factors such as the restricted range of motion of straight forceps and the impact of hand tremors on surgical precision. These challenges necessitate the development of more advanced techniques. The Da Vinci robotic surgical system plays a critical role in enhancing the precision of robotic surgeries. It provides a three-dimensional, ten-fold magnified view of the surgical area, promotes natural hand-eye coordination, filters hand tremors, and allows for greater freedom of movement with its articulated instruments. The benefits of the Da Vinci system have been proved in complex procedures such as D2 lymph node dissection for gastric cancer and lower mediastinal lymph node dissection. For example, during lower mediastinal lymph node dissection in adenocarcinoma of the gastroesophageal junction, the limited field of view of laparoscopic surgery restricts the use of linear instruments, whereas the flexibility of robotic surgery offers an advantage. Furthermore, peripancreatic lymph node clearance in radical gastric cancer surgery presents a challenge. LG is prone to causing pancreatic injury during dissection due to the fixed trocar positions and the rigidity of linear energy instruments, which can result in complications such as postoperative pancreatic fistulas and abdominal abscesses. The incidence of pancreatic fistulas after LG exceeds 5%, and higher amylase levels in drainage fluid suggest potential subclinical pancreatic injury. In contrast, robotic-assisted gastrectomy (RG) has evolved rapidly and offers advantages such as reduced pancreatic compression during dissection and a lower risk of thermal injury during lymph node removal. Retrospective studies suggest that RG is associated with less blood loss, shorter hospital stays, and improved lymph node dissection compared to LG. However, the evidence regarding the superiority of RG in terms of short-term outcomes remains controversial, as some prospective studies and meta-analyses have not confirmed its benefits. Prospective studies mainly focused on early gastric cancer, whereas the safety, efficacy, and cost-effectiveness of RG in advanced gastric cancer are still unclear.

Vascular coagulation is the key of minimally invasive surgery. In current robotic procedures, ultrasonic energy devices have been widely used. However, they lack flexibility and can generate high operating temperatures (up to 200°C), which risks thermal damage to surrounding tissues. Park et al. demonstrated that LG using bipolar energy devices resulted in lower postoperative C-reactive protein levels and reduced blood loss compared to ultrasonic scalpel use. The bipolar vascular closure system (Vessel Sealer Extend, VSE) is an advanced bipolar energy device with a fully articulated wrist joint, enabling 540° rotation and multi-directional access to vessels and target anatomical sites. The textured inner surface of the jaws enhances tissue grip, and it can coagulate vessels up to 7 mm in diameter with lower energy, minimizing thermal damage to adjacent structures. Retrospective studies have shown that robotic distal gastrectomy using VSE has earlier resumption of a semi-liquid diet (4.0 vs. 4.2 days, p=0.03) and a significantly lower incidence of postoperative intestinal obstruction (0% vs. 9.9%, p=0.03) compared to conventional laparoscopic surgery. The VSE has also demonstrated benefits in other surgical procedure. Yang et al. found that VSE use in robotic thyroidectomy reduced the frequency of camera cleaning compared to the Harmonic energy device (0.55 ± 0.51 vs. 1.93 ± 1.71, p<0.05). Additionally, a study comparing different robotic instrument combinations for adrenalectomy found that the VSE in combination with monopolar curved scissors offered the best performance. Based on these findings, the investigators believe that the VSE energy device could optimize RG, improving both safety and postoperative recovery.

There is a lack of prospective, multicenter, high-quality studies to verify the safety and recovery benefits associated with reduced thermal damage using this novel energy device. Therefore, the investigators propose a prospective, multicenter, observational cohort study to evaluate the safety, feasibility, and potential benefits of RG with the VSE energy device in the treatment of advanced gastric cancer. This study will assess postoperative recovery, inflammatory response, and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a, N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
* Preoperative abdominal enhanced CT and lung CT (or PET-CT) showed no distant metastasis
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) class I to III
* Written informed consent

Exclusion Criteria:

* Gastric multiple primary carcinoma or multiple primary cancer
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastric surgery (except ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection ) for gastric cancer)
* Preoperative gastric CT evaluation and chest and abdominal imaging evaluation were not performed before surgery, and the clinical stage of the tumor was not comprehensively evaluated
* Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
* History of other malignant disease within the past 5 years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within the past 6 months
* History of cerebrovascular accident within the past 6 months
* History of continuous systematic administration of corticosteroids within 1 month
* FEV1<50% of the predicted values
* Women during pregnancy or breast-feeding
* Severe mental disorder
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* Preoperative evaluation requires combined organ resection
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Primary gastric adenocarcinoma at the stage of cT2-4a, N-/+, M0.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall postoperative morbidity rates | Within 30 days after surgery
  Overall complication rates within 30 days after surgery in patients.

SECONDARY OUTCOMES:
comprehensive complication index, CCI | Within 30 days after surgery
  It was calculated according to the severity of surgical complications.
Intraoperative morbidity rates | Within 30 days after surgery
  The number of patients who received surgical treatment was used as the denominator, and the number of patients with intraoperative complications was used as the numerator.
Overall postoperative serious morbidity rates | Within 30 days after surgery
  According to the Clavien Dindo complication scoring system, IIIa and above were considered as severe complications, and when multiple complications occurred at the same time, the complication with the highest grade was considered.
Number of retrieved lymph nodes | Within 30 days after surgery
  The total number of harvested lymph nodes was confirmed by pathology.
Postoperative recovery | Within 30 days after surgery
  The recovery of patients after surgery, including physical and functional recovery, etc.
Postoperative prealbumin | 36 months
  Blood examination
Postoperative albumin | 36 months
  Blood examination
Inflammatory reponses | Within 30 days after surgery
  WBC, blood examination
Immune response | Within 30 days after surgery
  IL-6, blood examination
Immune response | Within 30 days after surgery
  IL-10, blood examination
Surgical costs | Within 30 days after surgery
  The cost of the patient's surgical treatment.
3-years disease free survival rates | Follow-up evaluations are performed up to 3 years postoperatively.
  The rate of 3-year disease free survival rates
3-year overall survival rates | Follow-up evaluations are performed up to 3 years postoperatively.
  The rate of 3-year overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes